CLINICAL TRIAL: NCT06141239
Title: Using 2D/3D Imaging to Analyze the Regeneration Rate of Autologous Bone During Alveolar Bone Preservation Surgery Using Periodontal Valves to Completely Cover Autologous Tooth Roots, Bone Substitutes, and Vitamin D3 Treatment
Brief Title: 2D/3D Imaging to Analyze the Regeneration Rate of Autologous Bone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsiang-Hsi Hong, Professor-level attending physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202102214A0
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Alveolar Ridge Preservation
MeSH Terms: interventions — Calcitriol; Bone Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- primary closure +Collagen plug +Bone graft (No Intervention): Placement of bone graft and collagen plug
- primary closure + Collagen plug +Bone graft +Vit.D3 (Experimental): Placement of bone graft, collagen plug and local administration of Vit.D3
  Interventions: Drug: Vit.D3; Other: bone graft
- primary closure +Collagen plug+Bone graft+Autologous Tooth Root (Experimental): Placement of bone graft, collagen plug and placement of autologous root slices
  Interventions: Procedure: Autologous Tooth Root; Other: bone graft
- primary closure +Collagen plug+Bone graft+Autologous Tooth Root+Vit.D3 (Experimental): Placement of bone graft, collagen plug and local administration of Vit.D3, and placement of autologous root slices
  Interventions: Procedure: Autologous Tooth Root; Drug: Vit.D3; Other: bone graft

INTERVENTIONS:
Procedure: Autologous Tooth Root — An autologous Tooth Root is made from one's own tooth root and covered in an extraction socket where bone graft is placed.
  Arms: primary closure +Collagen plug+Bone graft+Autologous Tooth Root; primary closure +Collagen plug+Bone graft+Autologous Tooth Root+Vit.D3
Drug: Vit.D3 — Local administration of Vit.D3, through the effect of Vit.D3 to explore whether it can help to accelerate the healing of tooth extraction cavity and the clinical effectiveness of bone regeneration
  Other Names: calcitriol
  Arms: primary closure + Collagen plug +Bone graft +Vit.D3; primary closure +Collagen plug+Bone graft+Autologous Tooth Root+Vit.D3
Other: bone graft — Selecting bone materials for alveolar ridge preservation according to treatment needs
  Other Names: BG
  Arms: primary closure + Collagen plug +Bone graft +Vit.D3; primary closure +Collagen plug+Bone graft+Autologous Tooth Root; primary closure +Collagen plug+Bone graft+Autologous Tooth Root+Vit.D3

SUMMARY:
Place a collagen plug (collagen plug) in the lower 2/3 to 1/2 of your tooth extraction site while giving you Vit. The extracted teeth are made into autogenous tooth root thin slices and covered in your tooth extraction cavity, and the skin flap raised by your flap surgery is used to cover the autologous tooth root cover to help the autologous tooth roots stabilize and heal the wound, which is different from traditional surgery. The difference in treatment lies in the local use of autogenous tooth root thin slices and Vit.D3. Collagen plug and Vit.D3 are already qualified medical materials and drugs on the market. However, there is no precedent for making thin autologous tooth root slices. will be a trial of a new medical technology that has not yet been used

DETAILED DESCRIPTION:
After tooth extraction, the shape of the alveolar bone will be changed. The ridge preservation method combined with the extraction socket sealing method has a significant clinical effect in preserving the vertical and horizontal directions of the alveolar bone ridge, and improves the predictability of the position of the dental bridge. and beautiful. Since there will be different bone formation rates in different locations of the extraction cavity, the literature shows that the bone formation rate is higher in the apical position of the extraction cavity, while the bone formation rate is lower in the coronal location. Therefore, the bone formation rate is 2/3~1/ under the extraction cavity. Insert the collagen plug at the 2 position and carry Vit.D3, and place appropriate bone material at the 1/3 position. If there is no bone material support, there will be a 50~60% chance that the autogenous root cover will fall off, but if all bone materials are placed at Under 3D imaging technology, it is impossible to clearly distinguish whether the image is the bone material itself or the formation of autogenous bone. Collagen plug uses its biocompatibility and absorbability and other biological properties to quickly stop bleeding and stabilize the clot in the wound, and has an impact on fibroblasts. It also has a chemotactic effect, accelerating the healing of extraction sockets, and can also promote the secretion of immature osteoid from the extracellular matrix. Vit.D3 can induce the differentiation of mesenchymal cells into osteoblasts and promote bone formation. Try to use these two Can the combination of biological materials and pharmaceuticals increase the bone formation rate? In addition, a cover made of autologous tooth root slices can be used for tooth extraction cavity sealing to prevent the bone material from being disturbed and damaged by the external environment. However, the autologous tooth root cover has a chance of falling off, so The skin flap opened by flap surgery is used to cover the autogenous tooth root cap, which strengthens the fixation and helps primary wound closure, reduces saliva contamination of bone graft materials, and accelerates wound healing. At the same time, it does not increase material costs or the patient's financial burden. Observe and track the treatment effect, and explore whether the shedding rate of autogenous root caps with and without valve coverage has an impact on alveolar ridge resorption. In addition, medical imaging technology is used to replace expensive and complicated biopsies, reduce the damage caused by biopsy to the structural integrity of the extraction socket, test whether there is new bone formation in the extraction socket, and integrate computer tomography and intraoral scan files, while observing the softness of the extraction socket. Hard tissue healing status.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign written subject consent
2. The tooth extraction socket is located in the anterior and posterior areas of the upper and lower jaws.
3. The area of the extraction socket (bone defect) in the mouth will need to be treated with artificial dental implants in the future.
4. The patient does not have systemic diseases (such as patients with hypertension, osteoporosis, bone-related diseases, kidney disease, thyroid and parathyroid diseases, etc.).

Exclusion Criteria:

1. Patients with potentially weakened healing abilities such as cancer, diabetes, bone infection, tuberculosis, anemia due to heme abnormalities or congenital immune deficiency, cellulitis, acute periodontal cyst, severe cusp disease (cyst size) >2mm2) or patients with dental and jaw lesions.
2. Women who are pregnant or breastfeeding.
3. Exclude heavy smokers or betel nut chewers who smoke more than one pack of cigarettes per day.
4. The bone defect in the extraction socket is severe and requires other bone regeneration surgeries (GBR), otherwise it will not be possible to have enough volume to provide artificial dental implants in the future.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
3D computed tomography data | At the 0th week and 12th~16th week of the experiment
  This experiment mainly used the relative position of the extraction socket and the adjacent tooth CEJ in CT images for height positioning and correction, and measured and compared the changes of the width and height of the bone ridge
  - Page 3 of 5 - and the shape and volume during the treatment. The Hu value of the adjacent dentin of the secondary CT was used as the standard and correction to measure and compare the change of the Hu value of the extraction socket during the treatment
periapical X-ray | 16 weeks after tooth extraction (before dental implants or other treatments)
  Take X-rays 16 weeks after tooth extraction (before dental implants or other treatments), record the width and height of the alveolar bone, and compare whether there is any difference in pixel values between the extraction socket and the adjacent non-extraction area, by calculating the number of pixels The difference in gray scale depth (i.e. density) of the image is determined by size to infer the formation of autogenous bone.
Intraoral scanner measurement data | At the 0th week and 12th~16th week of the experiment
  Follow-up observation and measurement: Intraoral photography scans were performed 0 weeks after tooth extraction/alveolar ridge preservation to record the appearance of soft tissues, including soft tissue thickness, buccal keratinized gingival width and thickness, and 16 weeks after surgery before dental implant surgery or other treatments. A second intraoral photography scan was performed to record the soft tissue condition again and compare the soft tissue wound healing evolution of the two tooth extraction cavities.
RFA measures implant stability (ISQ) | At the 16th~24th week of the experiment
  The implant stability was measured twice during the dental implant surgery at 16 to 24 weeks. The ISQ value of the 3.3mm diameter implant measured by Osstell Mentor was used as the standard ISQ value for correction. After the 3.3mm implant was removed, the matching funds would not be Then use a 3.3mm implant, and then measure the ISQ value of the implant (diameter 4.1 or 4.8mm) as the actual ISQ value of the initial stability of the implant. The implant repair will be made 3-4 months after the operation. Before implantation), measure the ISQ value of the second-stage stability of the implant to compare and analyze the changes in ISQ value of different implant groups and/or time points. Each subject followed this procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No